CLINICAL TRIAL: NCT06100575
Title: A Tool for Siblings and Children of Someone With Suicidal Thoughts and/or Behaviors: Evaluation.
Brief Title: Tool for Sibling and Children of Someone With Suicidal Thoughts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B6702023000493 - ONZ-2023-0335
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Website (www.mee-leven.be) (Experimental): Participants in this group (all participants) are asked to complete a questionnaire and then receive access to the website during three days, after which they were asked to complete another questionnaire.
  Interventions: Behavioral: Website (www.mee-leven.be)

INTERVENTIONS:
Behavioral: Website (www.mee-leven.be) — The tool is a website aimed siblings and children of someone who has suicidal thoughts and/or behaviors. The intended objectives of the tool are 1) to contribute to knowledge about suicide and health care options, 2) to increase perceived competences in dealing with suicidality of a family member, 3) to reduce perceived pressure and negative feelings such as hopelessness and 4) to be accessible and user-friendly.
  These objectives are achieved by providing the following content: 1) concerning the sibling/child themselves (primary objective) : information about the potential impact of having a suicidal family member, own needs, informal and formal (self) care, dealing with the suicidal family member, dealing with other family members 2) concerning the suicidal family member (Secondary objective): information about the suicidal process, signal recognition, how to provide support/create a safe environment for suicidal loved ones , help available for suicidal relatives

SUMMARY:
This study aims to investigate to what extent a website developed for siblings and children (16-25 years old) of someone with suicidal thoughts and/or behaviors is effective in improving perceived pressure, knowledge, attitudes, self-confidence and hopelessness. Moreover, it aims to examine how participants evaluate the website.

ELIGIBILITY:
Inclusion Criteria:

* Siblings and children of someone who has suicidal thoughts and/or behavior
* 16-25 years old
* Have access to internet
* Speak Dutch

Exclusion Criteria:

* /

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Changes in self-efficacy: Gatekeeper Self-Efficacy Scale (Takahashi et al., 2020) | Change from Baseline (before intervention) to post-test (after 3 days of access to website)
  The Gatekeeper Self-Efficacy Scale is a 9-item self-report scale to be scored on a 7-point Likert scale (1= not at all to 5 = Extremely) to measure participants' self efficacy in dealing with suicidal individuals. Higher scores indicate higher self-efficacy.

SECONDARY OUTCOMES:
Changes in perceived pressure: Perceived pressure informal care ('Ervaren druk informele zorg', Pot et al., 1995) | Change from Baseline (before intervention) to post-test (after 3 days of access to website)
  The Perceived pressure informal care ('Ervaren druk informele zorg', Pot et al., 1995) scale is a 9-item self-report scale. Participants rate items to be applicable to them with the options: 'No!', 'No', 'More or less', 'Yes', 'Yes!', where 'No' and 'No!' are scored as 0 and the other options as 1. Total scores of 0-3 indicate little pressure, 4-6 moderate and 7-9 a lot.
Changes in attitudes: 5 subscales of Attitudes Towards Suicide Scale (Rensberg & Jacobson, 2003; De Clerck et al., 2006) | Change from Baseline (before intervention) to post-test (after 3 days of access to website)
  The ATTS is a 37-item to be scored on a 5-point Likert scale (1= disagree completely to 5 = agree completely) to measure participants' attitudes towards suicide. The included subscales in this study are: incomprehensibility, non-communication, preventability, tabooing, preparedness to prevent
Changes in hopelessness: Beck Hopelessness Scale (4-item version; Beck et al., 1974; Aish & Wasserman, 2001) and self-developed questionnaire | Change from Baseline (before intervention) to post-test (after 3 days of access to website)
  The BHS A 4-item self-report questionnaire to measure hopelessness in adolescents and adults. Each item is rated as 'true' (score = 1) or 'false' (score = 0) for them over the past week, resulting in a total score ranging from 0 to 4, with higher scores indicating higher levels of hopelessness.
  Self-developed questionnaire: 4-item self-report questionnaire to measure hopelessness in relation to the loved one, based on the BHS 4-item version. Each item is rated as 'true' (score = 1) or 'false' (score = 0) for them over the past week, resulting in a total score ranging from 0 to 4, with higher scores indicating higher levels of hopelessness in relation to the loved one.
Changes in self-care and awareness | Change from Baseline (before intervention) to post-test (after 3 days of access to website)
  Self-developed questionnaire consisting of 5 statements to be rated on a 5-point Likert scale, with 1=strongly disagree and 5=strongly agree. Higher scores indicate higher levels of self-care and awareness.
Evaluation of the website | post-test (after 3 days of access to website)
  18 statements about the content, structure and effect of the website to be rated on a 5-point Likert scale (1= strongly disagree, 5= strongly agree) 4 open questions: "Which part of the website benefited you the most and why?"; "Which part of the website benefited you the least and why?"; "What can be improved on the website?" "Would you like to say anything else about the website?" Participants were asked to rate the website on a scale of 1-10

OTHER OUTCOMES:
Socio-demographic characteristics | Baseline
  age (continuous), gender (man, woman, other), previous health care (yes/no; categories 'professional healthcare provider', 'suicide prevention helpline', 'other'), needed health care (yes/no)
Characteristics of the suicidal family member | Baseline
  relationship to participant (parent, sibling), previous thoughts and/or attempts (never, sometimes, regularly, n/a; as estimated by the participant), age (continuous), gender (man, woman, other)

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Portzky, Phd, Principal Investigator — University Ghent
Locations (1):
- Flemish Centre of Expertise in Suicide Prevention, Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No